CLINICAL TRIAL: NCT00048542
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Efficacy, and Pharmacokinetics of the Human Anti-TNF Monoclonal Antibody Adalimumab in Children With Polyarticular Juvenile Idiopathic Arthritis
Brief Title: Study of Human Anti-TNF Monoclonal Antibody Adalimumab in Children With Polyarticular Juvenile Idiopathic Arthritis (JIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DE038
Record Dates: First submitted 2002-11-01; First posted 2002-11-05 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Arthritis, Juvenile Idiopathic
Keywords: Polyarticular Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Double-Blind Adalimumab + MTX (Experimental): Subjects who were inadequate responders to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase received adalimumab plus concomitant MTX during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
  Interventions: Biological: Double-Blind Adalimumab/Placebo + MTX
- Double-Blind Placebo + MTX (Placebo Comparator): Subjects who were inadequate responders to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase received placebo plus concomitant MTX during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
  Interventions: Biological: Double-Blind Adalimumab/Placebo + MTX
- Double-Blind Adalimumab (Experimental): Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received adalimumab, but no concomitant MTX treatment, during the Double-Blind Phase.
  Interventions: Biological: Double-Blind Adalimumab/Placebo
- Double-Blind Placebo (Placebo Comparator): Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received placebo, but no concomitant MTX treatment, during the Double-Blind Phase.
  Interventions: Biological: Double-Blind Adalimumab/Placebo
- OLE BSA Adalimumab + MTX (Experimental): All subjects received subcutaneous injections of 24 mg adalimumab per square meter of body surface area (BSA) up to a maximum of 40 mg total body dose every other week (eow), concomitantly with MTX treatment, during the Open-Label Extension (OLE) BSA Phase of the study.
  Interventions: Drug: OLE BSA Adalimumab +/- MTX
- OLE BSA Adalimumab (Experimental): All subjects received subcutaneous injections of 24 mg adalimumab per square meter of body surface area (BSA) up to a maximum of 40 mg total body dose every other week (eow), but not MTX treatment, during the Open-Label Extension (OLE) BSA Phase of the study.
  Interventions: Drug: OLE BSA Adalimumab +/- MTX
- OLE FD Adalimumab + MTX (Experimental): Subjects received adalimumab concomitantly with MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study in which only body weight (not BSA) determined dosing; subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
  Interventions: Drug: OLE FD Adalimumab +/- MTX
- OLE FD Adalimumab (Experimental): Subjects received placebo without concomitant MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study in which only body weight (not BSA) determined dosing; subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
  Interventions: Drug: OLE FD Adalimumab +/- MTX

INTERVENTIONS:
Biological: Double-Blind Adalimumab/Placebo + MTX — Subcutaneous injection of 24 mg adalimumab or placebo per square meter of body surface area (BSA) every other week (eow) concomitantly with MTX treatment for 32 weeks during the Double-Blind phase. Total body dose of adalimumab was not to exceed 40 mg.
  Other Names: ABT-D2E7; Humira
  Arms: Double-Blind Adalimumab + MTX; Double-Blind Placebo + MTX
Biological: Double-Blind Adalimumab/Placebo — Subcutaneous injection of 24 mg adalimumab or placebo per square meter of body surface area (BSA) every other week (eow) without MTX treatment for 32 weeks during the Double-Blind Phase. Total body dose of adalimumab was not to exceed 40 mg.
  Other Names: ABT-D2E7; Humira
  Arms: Double-Blind Adalimumab; Double-Blind Placebo
Drug: OLE BSA Adalimumab +/- MTX — Comparison of subcutaneous injection of 24 mg adalimumab per square meter of body surface area (BSA) every other week (eow) either with or without concomitant MTX treatment for a minimum of 44 weeks (up to a maximum of 136 weeks) during the Open-Label Extension BSA Phase.
  Other Names: ABT-D2E7; Humira
  Arms: OLE BSA Adalimumab; OLE BSA Adalimumab + MTX
Drug: OLE FD Adalimumab +/- MTX — Comparison of adalimumab administered subcutaneously every other week (eow) either with or without concomitant MTX treatment for up to 224 weeks during the Open-Label Extension Fixed Dose (FD) Phase.
  Other Names: ABT-D2E7; Humira
  Arms: OLE FD Adalimumab; OLE FD Adalimumab + MTX

SUMMARY:
This is a multicenter, Phase 3 randomized, placebo-controlled study designed to evaluate adalimumab in children 4 to 17 years old with polyarticular juvenile idiopathic arthritis (JIA) who are either methotrexate (MTX) treated or non-MTX treated.

DETAILED DESCRIPTION:
The study design for this clinical trial was chosen to evaluate adalimumab in subjects who were either methotrexate (MTX)-naive or had been withdrawn from MTX at least 2 weeks prior to study drug administration (non-MTX stratum) or were inadequate responders to MTX and continued MTX treatment (MTX stratum). The study consisted of 4 phases: a 16-week Open-label Lead-in (OL LI), a 32-week Double-blind (DB) phase, an up to 136-week Open-label Extension Body Surface Area (OLE BSA) phase, and an up to 224-week OLE Fixed Dose (FD) phase. All subjects who met entry criteria were enrolled into one of the appropriate strata and received adalimumab (plus concomitant MTX in the MTX stratum) in the 16 week OL LI phase of the study. All subjects who responded to adalimumab during the OL LI phase were to be enrolled in the DB phase of the study and randomized to receive adalimumab (plus concomitant MTX in the MTX stratum) or placebo (plus concomitant MTX in the MTX stratum). Subjects in the DB phase received either adalimumab (24 mg/m2 BSA up to a maximum of 40 mg total body dose) or placebo subcutaneously (SC) administered every other week (eow). Adalimumab or placebo was administered for an additional 32 weeks or until flare of disease (based on PedACR30 response criteria = a worsening of 30% or more in 3 of the 6 response variables (Parent's global assessment of subject's overall well-being by visual analog scale [VAS], Physician's global assessment [PhGA] of subject's disease severity by VAS, number of active joints [joints with swelling not due to deformity or joints with limitation of passive motion (LOM)], pain, tenderness, or both, number of joints with LOM, Childhood Health Assessment Questionnaire [CHAQ], and CRP levels), a minimum of 2 active joints, and no more than 1 indicator improving by 30% or more), whichever occurred earlier. For subjects who did not have a disease flare, the DB phase was completed at Week 48. Subjects who experienced disease flare during the DB phase or subjects who completed 48 weeks of the study were given the option to receive adalimumab for up to a minimum of 44 weeks (up to a maximum of 136 weeks) in the OLE BSA phase before being eligible to switch to the OLE FD phase. In this phase, subjects received OL adalimumab (24 mg/m2 BSA up to a maximum of 40 mg total body dose SC eow). All subjects who completed at least 44 weeks of OLE BSA treatment were given the opportunity to continue into the OLE FD phase for up to 224 weeks of additional adalimumab exposure. In this phase, subjects weighing less than 30 kg were treated with a fixed dose of 20 mg of adalimumab SC eow. Subjects weighing 30 kg or more were treated with a fixed dose of 40 mg of adalimumab SC eow.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of polyarticular juvenile idiopathic arthritis (JIA) age 4 to 17 by the American College of Rheumatology (ACR) criteria. Disease onset may have been systemic, polyarticular, or pauciarticular. If the disease was systemic onset, then the subjects must be free of any systemic JIA manifestations for at least 3 months before the time of qualification.
* At the time of study screening, the subject must have continuing active disease defined as >= 5 swollen joints and >= 3 joints with limitation of motion (LOM). These joints are not mutually exclusive.
* Subjects may be either naïve to MTX, inadequate responders to MTX, or intolerant to MTX. Intolerance to MTX will be defined by the subject's physician. The MTX must be maintained at a dose of at least 10 mg/m2 body surface area/week for a minimum of 3 months, prior to screening.
* Duration of disease is not limited, but must have been long enough for a subject to have been given an adequate trial of nonsteroidal anti-inflammatory drugs (NSAIDs).
* Have not received other disease-modifying anti-rheumatic drugs (DMARDs) including penicillamine, hydroxychloroquine, sulfasalazine, oral or injectable gold, cyclosporin; or intravenous immunoglobulin (IV Ig); or cytotoxic agents, for at least 4 weeks prior to receiving 1st dose of study drug. Subjects currently on one or more of these DMARDs must demonstrate active disease (defined above) prior to a minimum 4 weeks (28 days) washout of all DMARDs.
* Subjects who are refractory to MTX after 3 months of treatment must demonstrate active disease (defined above) prior to enrollment in the open-label part of the trial.
* Have not received an intra-articular glucocorticoid injection within 4 weeks (28 days) prior to enrollment into the study.
* Have good venous access and stable hematocrit >= 24%.
* All sexually active male and female study participants must be practicing adequate contraception. Post-pubertal females must have a negative serum pregnancy test no greater than 10 days prior to the first dose of study drug.
* Parent or guardian has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject's parent or legal guardian has had the opportunity to ask questions.

Exclusion Criteria:

* Pregnant or nursing female.
* Functional class IV by ACR criteria.
* Laboratory parameters outside limits established in the protocol.
* Medical history, medical condition, or previous treatment not allowed by the protocol.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2002-09; Primary Completion 2005-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, M.D., Ph.D., Study Director — Abbott
Locations (31):
- United States (15):
  - Site Ref # / Investigator 45524, Birmingham, Alabama
  - Site Reference ID/Investigator# 2235, Los Angeles, California
  - Site Reference ID/Investigator# 642, Stanford, California
  - Site Reference ID/Investigator# 638, Delray Beach, Florida
  - Site Ref # / Investigator 45543, St. Petersburg, Florida
  - Site Reference ID/Investigator# 640, Chicago, Illinois
  - Site Reference ID/Investigator# 644, Kansas City, Kansas
  - Site Reference ID/Investigator# 641, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 645, Omaha, Nebraska
  - Site Reference ID/Investigator# 2501, Livingston, New Jersey
  - Site Ref # / Investigator 45542, New Hyde Park, New York
  - Site Ref # / Investigator 45544, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 386, Columbus, Ohio
  - Site Ref # / Investigator 45525, Salt Lake City, Utah
  - Site Reference ID/Investigator# 406, Norfolk, Virginia
- Belgium (2):
  - Site Reference ID/Investigator# 621, Ghent
  - Site Reference ID/Investigator# 2538, Leuven
- Czechia (2):
  - Site Reference ID/Investigator# 519, Prague
  - Site Reference ID/Investigator# 518, Prague
- France (2):
  - Site Reference ID/Investigator# 45545, Marseille
  - Site Reference ID/Investigator# 516, Paris
- Germany (5):
  - Site Reference ID/Investigator# 627, Berlin
  - Site Reference ID/Investigator# 625, Bremen
  - Site Ref # / Investigator 45522, Garmisch-Partenkirchen
  - Site Reference ID/Investigator# 628, Halle
  - Site Reference ID/Investigator# 622, Hamburg
- Italy (2):
  - Site Reference ID/Investigator# 631, Genoa
  - Site Reference ID/Investigator# 636, Milan
- Slovakia (2):
  - Site Ref # / Investigator 45523, Košice
  - Site Reference ID/Investigator# 3425, Piešťany
- Site Reference ID/Investigator# 3713, Madrid, Spain

REFERENCES:
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- [Derived] Lovell DJ, Ruperto N, Goodman S, Reiff A, Jung L, Jarosova K, Nemcova D, Mouy R, Sandborg C, Bohnsack J, Elewaut D, Foeldvari I, Gerloni V, Rovensky J, Minden K, Vehe RK, Weiner LW, Horneff G, Huppertz HI, Olson NY, Medich JR, Carcereri-De-Prati R, McIlraith MJ, Giannini EH, Martini A; Pediatric Rheumatology Collaborative Study Group; Pediatric Rheumatology International Trials Organisation. Adalimumab with or without methotrexate in juvenile rheumatoid arthritis. N Engl J Med. 2008 Aug 21;359(8):810-20. doi: 10.1056/NEJMoa0706290. PMID 18716298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 31 sites between 19 September 2002 and 13 January 2005.
Pre-assignment Details: A total of 171 participants entered the Open-Label Lead-In (OL-LI) phase and received adalimumab. Of these 171 participants, 160 participants completed the OL-LI phase, and 133 participants entered the 32-week Double-Blind Phase (75 in the MTX stratum; 58 in the non-MTX stratum) and were randomized to adalimumab or placebo.
Groups:
- Double-Blind Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received adalimumab (24 mg/square meter of body surface area [BSA], up to a maximum of 40 mg total body dose administered subcutaneously every other week) plus concomitant MTX treatment during the Double-Blind Phase of the study. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
- Double-Blind Placebo + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received placebo (24 mg/square meter of body surface area [BSA], up to a maximum of 40 mg total body dose administered subcutaneously every other week) plus concomitant MTX treatment during the Double-Blind Phase of the study.
  MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
- Double-Blind Adalimumab: Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received adalimumab (24 mg/square meter of body surface area [BSA], up to a maximum of 40 mg total body dose administered subcutaneously every other week), but no concomitant MTX treatment, during the Double-Blind Phase of the study.
- Double-Blind Placebo: Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received placebo (24 mg/square meter of body surface area [BSA], up to a maximum of 40 mg total body dose, administered subcutaneously every other week), but no concomitant MTX treatment, during the Double-Blind Phase of the study.
- Open-Label Extension BSA Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum received subcutaneous injections of 24 mg adalimumab per square meter of body surface area (BSA) up to a maximum of 40 mg total body dose every other week (eow) concomitantly with MTX treatment during the Open-Label Extension BSA Phase of the study.
- Open-Label Extension BSA Adalimumab: Subjects in the non-methotrexate (MTX) stratum received adalimumab (24 mg/square meter of body surface area [BSA], up to a maximum of 40 mg total body dose SC eow) without concomitant MTX treatment during the Open-Label Extension BSA Phase.
- Open-Label Extension FD Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum received adalimumab concomitantly with MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study in which only body weight (not BSA) determined dosing. Subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
- Open-Label Extension FD Adalimumab: Subjects in the non-methotrexate (MTX) stratum received adalimumab without concomitant MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study in which body weight (not BSA) determined dosing. Subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
Period: Double-Blind Phase
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX | Double-Blind Adalimumab | Double-Blind Placebo | Open-Label Extension BSA Adalimumab + MTX | Open-Label Extension BSA Adalimumab | Open-Label Extension FD Adalimumab + MTX | Open-Label Extension FD Adalimumab
Started | 38 (For all groups, started indicates when the subjects entered the double-blind treatment phase.) | 37 | 30 | 28 | 0 | 0 | 0 | 0
Completed | 35 | 36 | 29 | 28 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor request or decision | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized in error | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Extension BSA Phase
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX | Double-Blind Adalimumab | Double-Blind Placebo | Open-Label Extension BSA Adalimumab + MTX | Open-Label Extension BSA Adalimumab | Open-Label Extension FD Adalimumab + MTX | Open-Label Extension FD Adalimumab
Started | 0 | 0 | 0 | 0 | 71 | 57 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 59 | 47 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 10 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 6 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor request or decision | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Period: Open-Label Extension Fixed Dose Phase
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX | Double-Blind Adalimumab | Double-Blind Placebo | Open-Label Extension BSA Adalimumab + MTX | Open-Label Extension BSA Adalimumab | Open-Label Extension FD Adalimumab + MTX | Open-Label Extension FD Adalimumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 59 | 47
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Sponsor request or decision | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX | Double-Blind Adalimumab | Double-Blind Placebo | Total
Number analyzed (Participants) | 38 | 37 | 30 | 28 | 133
Age Continuous [Mean (Standard Deviation); unit: years] — Age for participants in the Double-Blind Phase only.
  years | 11.7 (3.29) | 10.8 (3.36) | 11.1 (4.13) | 11.3 (3.77) | 11.2 (3.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Numbers represent participants in the Double-Blind Phase only.
  Participants
    Female | 30 | 30 | 23 | 20 | 103
    Male | 8 | 7 | 7 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in the Non-MTX Stratum With Disease Flare During the Double-Blind Phase
Description: The primary efficacy endpoint was the number of adalimumab-treated subjects in the non-MTX stratum with disease flare during the Double-Blind Phase compared with the number of placebo-treated subjects in the non-MTX stratum with disease flare during the double-blind phase. Subjects met the criteria for disease flare if they had 1) >= 30% worsening in at least 3 of the 6 Juvenile Rheumatoid Arthritis (JRA) core set criteria and a minimum of 2 active joints, and 2) >= 30% improvement in not more than 1 of the 6 JRA core set criteria.
Time Frame: Week 16 to Week 48 (32 weeks)
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug, in the non-MTX stratum. Missing values were treated as disease flare.
Measure: Number; unit: Participants
Groups:
- Double-Blind Adalimumab: Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received adalimumab (24 mg/square meter of body surface area [BSA], not to exceed 40 mg, every other week), but no concomitant MTX treatment, during the Double-Blind Phase of the study.
- Double-Blind Placebo: Subjects in the non-methotrexate (MTX) stratum who were either naïve to MTX or withdrawn from MTX at least 2 weeks prior to study drug administration, and were adalimumab responders during the OL-LI phase, received placebo (24 mg/square meter of body surface area [BSA], not to exceed 40 mg, every other week), but no concomitant MTX treatment, during the Double-Blind Phase of the study.
Arm/Group | Double-Blind Adalimumab | Double-Blind Placebo
Number analyzed (Participants) | 30 | 28
Participants | 13 | 20
Statistical Analysis 1: Comparison: Double-Blind Adalimumab vs Double-Blind Placebo; The study was sized to detect a difference in the proportion of subjects (40%) between placebo and the active adalimumab dose group who would experience disease flare assuming a placebo rate of 70% vs. a rate of 30% in the active group. Assuming a binomial distribution, an alpha of 0.05, 80% power, two-sided test, and an initial monotherapy responder rate of 70%, a minimum of 29 subjects were needed per treatment group within the appropriate strata; Test type: Superiority or Other; p = 0.031, Chi-square test

2. Secondary Outcome: Number of Subjects Meeting Pediatric American College of Rheumatology 30% (PedACR30) Response Criteria at the End of the Open-Label Lead-In Phase
Description: Responders met the following criteria: >= 30% improvement in >= 3 of 6 JRA core set criteria, and >= 30% worsening in not more than 1 JRA criterion, compared with the open-label baseline. JRA core set criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with limitation of motion [LOM] and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein.
Time Frame: Week 16
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug. Missing values were treated as non-responders.
Measure: Number; unit: Participants
Groups:
- Adalimumab + MTX: Subjects received methotrexate (MTX) plus open-label adalimumab (24 mg/square meter up to a maximum of 40 mg total body dose by body surface area [BSA] administered subcutaneously [SC] every other week [eow]) during the Open-Label Lead-In (OL-LI) Phase of the study.
- Adalimumab: Subjects received open-label adalimumab (24 mg/square meter up to a maximum of 40 mg total body dose by body surface area [BSA] administered subcutaneously [SC] every other week [eow]), but no methotrexate (MTX), during the Open-Label Lead-In (OL-LI) Phase of the study.
Arm/Group | Adalimumab + MTX | Adalimumab
Number analyzed (Participants) | 85 | 86
Participants | 80 | 64

3. Secondary Outcome: Number of Subjects in the MTX Stratum With Disease Flare During the Double-Blind Phase
Description: Subjects met criteria for disease flare if they had >= 30% worsening in at least 3 of 6 JRA core set criteria and a minimum of 2 active joints, and >= 30% improvement in not more than 1 JRA criterion. JRA core set criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with LOM and with pain, tenderness or both); number of joints with LOM; physical function of Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein.
Time Frame: Week 16 to Week 48 (32 Weeks)
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug, in the MTX stratum. Missing values were treated as disease flare.
Measure: Number; unit: Participants
Groups:
- Double-Blind Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received adalimumab plus concomitant MTX during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
- Double-Blind Placebo + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received placebo plus concomitant MTX during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX
Number analyzed (Participants) | 38 | 37
Participants | 14 | 24
Statistical Analysis 1: Comparison: Double-Blind Adalimumab + MTX vs Double-Blind Placebo + MTX; Test type: Superiority or Other; p = 0.015, Chi-square test

4. Secondary Outcome: Time to Onset of Disease Flare During the Double-Blind Phase in Subjects in the Non-MTX Stratum
Description: A log rank test was performed and the Kaplan-Meier curve for time to disease flare from double-blind baseline (Week 16) to Week 48 was generated. Disease flare was defined as a >= 30% worsening in at least 3 of 6 JRA core set criteria and a minimum of 2 active joints, and >= 30% improvement in not more than 1 JRA criterion. The percentage of subjects without disease flare at each time point is presented.
Time Frame: Week 16 to Week 48 (32 weeks)
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug, in the non-MTX stratum.
Measure: Number; unit: Percent participants w/o disease flare
Arm/Group | Double-Blind Adalimumab | Double-Blind Placebo
Number analyzed (Participants) | 30 | 28
Percent participants w/o disease flare
  Week 20 | 90.0 | 78.6
  Week 24 | 83.3 | 64.3
  Week 28 | 80.0 | 60.7
  Week 32 | 70.0 | 46.4
  Week 36 | 66.7 | 46.4
  Week 40 | 60.0 | 39.3
  Week 44 | 60.0 | 32.1
  Week 48 | 56.7 | 28.6
Statistical Analysis 1: Comparison: Double-Blind Adalimumab vs Double-Blind Placebo; Test type: Superiority or Other; p = 0.029, Log Rank

5. Secondary Outcome: Time to Onset of Disease Flare During the Double-Blind Phase in Subjects in the MTX Stratum
Description: as for outcome 4
Time Frame: Week 16 to Week 48 (32 weeks)
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug, in the MTX stratum.
Measure: Number; unit: Percent participants w/o disease flare
Groups:
- Double-Blind Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received adalimumab (24 mg per square meter of body surface area [BSA] every other week [eow]) plus concomitant MTX treatment during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
- Double-Blind Placebo + MTX: Subjects in the methotrexate (MTX) stratum, who had an inadequate response to MTX and were adalimumab responders during the Open-Label Lead-In (OL-LI) phase, received placebo (24 mg per square meter of body surface area [BSA] every other week [eow]) plus concomitant MTX treatment during the Double-Blind Phase. MTX-treated inadequate responders must have had active disease on MTX treatment for at least 3 months prior to screening.
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX
Number analyzed (Participants) | 38 | 37
Percent participants w/o disease flare
  Week 20 | 86.8 | 83.8
  Week 24 | 78.9 | 70.3
  Week 28 | 68.4 | 59.5
  Week 32 | 68.4 | 56.8
  Week 36 | 63.2 | 48.6
  Week 40 | 63.2 | 45.9
  Week 44 | 63.2 | 43.2
  Week 48 | 63.2 | 35.1
Statistical Analysis 1: Comparison: Double-Blind Adalimumab + MTX vs Double-Blind Placebo + MTX; Test type: Superiority or Other; p = 0.031, Log Rank

6. Secondary Outcome: Number of Subjects Meeting PedACR30 Response Criteria at the End of the Double-Blind Phase
Description: Responders met the following criteria: >= 30% improvement in >= 3 of 6 JIA core set criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with the OL baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with LOM and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. All core criteria are included in PedACR criteria.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Adalimumab: Subjects received adalimumab during the open-label lead-in phase and during the double-blind phase.
- Placebo: Subjects received adalimumab during the open-label lead-in phase and placebo during the double-blind phase.
- Adalimumab + MTX: Subjects received adalimumab plus MTX during the open-label lead-in phase and adalimumab plus MTX during the double-blind phase.
- Placebo + MTX: Subjects received adalimumab plus MTX during the open-label lead-in phase and placebo plus MTX during the double-blind phase.
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 30 | 28 | 38 | 37
Participants | 17 | 9 | 24 | 14
Statistical Analysis 1: Comparison: Adalimumab vs Placebo; Test type: Superiority or Other; p = 0.061, Pearson's Chi-square test
Statistical Analysis 2: Comparison: Adalimumab + MTX vs Placebo + MTX; Test type: Superiority or Other; p = 0.028, Pearson's Chi-square test

7. Secondary Outcome: Number of Subjects Meeting PedACR50 Response Criteria at the End of the Double-Blind Phase
Description: Responders met the following criteria: >= 50% improvement in >= 3 of 6 JIA core set criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with the OL baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with LOM and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. All core variables are included in PedACR criteria.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Adalimumab: Subjects received adalimumab during open-label lead-in phase and during the double-blind phase.
- Adalimumab + MTX: Subjects received adalimumab plus MTX during the open-label lead-in phase and adalimumab plus MTX double-blind phase.
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 30 | 28 | 38 | 37
Participants | 16 | 9 | 24 | 14
Statistical Analysis 1: Comparison: Adalimumab vs Placebo; Test type: Superiority or Other; p = 0.103, Pearson's Chi-square test
Statistical Analysis 2: Comparison: Adalimumab + MTX vs Placebo + MTX; Test type: Superiority or Other; p = 0.028, Pearson's Chi-square test

8. Secondary Outcome: Number of Subjects Meeting PedACR70 Response Criteria at the End of the Double-Blind Phase
Description: Responders met the following criteria: >= 70% improvement in >= 3 of 6 JIA core set criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with the OL baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with LOM and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. All core variables are included in PedACR criteria.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 30 | 28 | 38 | 37
Participants | 14 | 8 | 24 | 10
Statistical Analysis 1: Comparison: Adalimumab vs Placebo; Test type: Superiority or Other; p = 0.156, Pearson's Chi-square test
Statistical Analysis 2: Comparison: Adalimumab + MTX vs Placebo + MTX; Test type: Superiority or Other; p = 0.002, Pearson's Chi-square test

9. Secondary Outcome: Mean Change From Baseline in Physician's Global Assessment of Disease Activity at Week 48 of the Double-Blind Phase
Description: A 100 mm horizontal visual analog scale (VAS) was used to assess the Physician Global Assessment of Disease Activity. The left end of the VAS scale (0 mm) signified the absence of symptoms and the right end (100 mm) maximum disease activity. The mean change from open-label baseline to Week 48 was determined. Negative mean changes indicated improvement.
Time Frame: Baseline and Week 48
Population: All subjects in the intent-to-treat population, defined as all subjects who were randomized and who received at least a single administration of study drug, who completed Week 48. Observed data of subjects who remained in the study at Week 48 were analyzed.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 17 | 9 | 24 | 15
Units on a scale | -52.06 (3.713) | -38.73 (6.554) | -48.50 (3.890) | -38.73 (6.554)

10. Secondary Outcome: Mean Change From Baseline in Parent's/Patient's Global Assessment of Disease Activity at Week 48 of the Double-Blind Phase
Description: A 100 mm horizontal visual analog scale (VAS) was used to assess the Parent's/Patient's Global Assessment of Disease Activity. The left end of the VAS (0 mm) signified the absence of symptoms and the right end (100 mm) maximum disease activity. The mean change from open-label baseline to Week 48 was determined. Negative mean changes indicated improvement.
Time Frame: Baseline and Week 48
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 17 | 9 | 24 | 15
Units on a scale | -41.53 (5.562) | -50.56 (6.129) | -36.42 (5.177) | -26.87 (5.644)

11. Secondary Outcome: Mean Change From Baseline in C-Reactive Protein Levels at Week 48 of the Double-Blind Phase
Description: Serum levels of C-reactive protein (CRP) were measured at screening (open-label baseline) and at Week 48. Negative mean changes in CRP from open-label baseline to Week 48 indicated improvement.
Time Frame: Baseline and Week 48
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Adalimumab | Placebo | Adalimumab + MTX | Placebo + MTX
Number analyzed (Participants) | 17 | 9 | 24 | 15
mg/dL | -1.79 (0.803) | -3.91 (2.000) | -1.71 (0.529) | -0.10 (0.333)

12. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Baseline of the Open-Label Extension Body Surface Area Phase
Description: Responders met the following criteria: >= 30%/50%/70% improvement in >= 3 of 6 JIA core criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with OL baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; # of active joints (joints with swelling or with LOM and with pain, tenderness or both); # of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. All core assessments are included in PedACR criteria.
Time Frame: Open-Label Lead-In Phase Baseline
Population: The ITT population was used for analysis in the Open-Label Extension Body Surface Area phase.
Measure: Number; unit: Participants
Groups:
- OLE BSA Adalimumab + MTX: Subjects received adalimumab and concomitant MTX during the Open-Label Extension body surface area (BSA) phase. Subjects received OL adalimumab (24 mg/m2 BSA up to a maximum of 40 mg total body dose subcutaneously (SC) every other week (eow).
- OLE BSA Adalimumab: Subjects received adalimumab, but not concomitant MTX, during the Open-Label Extension body surface area (BSA) phase. Subjects received OL adalimumab (24 mg/m2 BSA up to a maximum of 40 mg total body dose subcutaneously (SC) every other week (eow).
Arm/Group | OLE BSA Adalimumab + MTX | OLE BSA Adalimumab
Number analyzed (Participants) | 67 | 53
Participants
  PedACR30 Baseline | 55 | 46
  PedACR50 Baseline | 47 | 41
  PedACR70 Baseline | 35 | 30

13. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Week 56 of the Open-Label Extension Body Surface Area Phase
Description: as for outcome 12
Time Frame: Week 56
Population: The ITT population was used for analysis in the Open-Label Extension Body Surface Area phase.
Measure: Number; unit: Participants
Arm/Group | OLE BSA Adalimumab + MTX | OLE BSA Adalimumab
Number analyzed (Participants) | 55 | 41
Participants
  PedACR30 Week 56 | 50 | 40
  PedACR50 Week 56 | 49 | 40
  PedACR70 Week 56 | 43 | 35

14. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Week 104 of the Open-Label Extension Body Surface Area Phase
Description: as for outcome 12
Time Frame: Week 104
Population: The ITT population was used for analysis in the Open-Label Extension Body Surface Area phase.
Measure: Number; unit: Participants
Arm/Group | OLE BSA Adalimumab + MTX | OLE BSA Adalimumab
Number analyzed (Participants) | 19 | 17
Participants
  PedACR30 Week 104 | 18 | 16
  PedACR50 Week 104 | 16 | 16
  PedACR70 Week 104 | 14 | 14

15. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Baseline of the Open-Label Extension Fixed Dose Phase
Description: Responders met the following criteria: >= 30%/50%/70% improvement in >= 3 of 6 JIA core criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with OL-LI baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; # of active joints (joints with swelling or with LOM and with pain, tenderness or both); # of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. All core assessments are included in PedACR criteria.
Time Frame: Baseline
Population: The ITT population was used for analysis in the Open-Label Extension Fixed Dose phase.
Measure: Number; unit: Participants
Groups:
- OLE FD Adalimumab + MTX: Subjects received adalimumab and concomitant MTX during the Open-Label Extension fixed dose phase. Subjects weighing less than 30 kg were dosed with 20 mg of adalimumab subcutaneously (SC) every other week (eow). Subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
- OLE FD Adalimumab: Subjects received adalimumab, but not concomitant MTX, during the Open-Label Extension Fixed Dose phase. Subjects weighing less than 30 kg were dosed with 20 mg of adalimumab subcutaneously (SC) every other week (eow). Subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 53 | 45
Participants
  PedACR30 OLE FD Baseline | 53 | 44
  PedACR50 OLE FD Baseline | 50 | 43
  PedACR70 OLE FD Baseline | 46 | 40

16. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Week 48 of the Open-Label Extension Fixed Dose Phase
Description: as for outcome 15
Time Frame: Week 48
Population: The ITT population was used for analysis in the Open-Label Extension Fixed Dose phase.
Measure: Number; unit: Participants
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 51 | 40
Participants
  PedACR30 Week 48 | 47 | 40
  PedACR50 Week 48 | 47 | 39
  PedACR70 Week 48 | 44 | 38

17. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at Week 112 of the Open-Label Extension Fixed Dose Phase
Description: as for outcome 12
Time Frame: Week 112
Population: The ITT population was used for analysis in the Open-Label Extension Fixed Dose phase.
Measure: Number; unit: Participants
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 41 | 31
Participants
  PedACR30 Week 112 | 39 | 31
  PedACR50 Week 112 | 39 | 30
  PedACR70 Week 112 | 34 | 29

18. Secondary Outcome: Number of Subjects Meeting PedACR30/50/70 Response Criteria at the Final Visit (up to 224 Weeks) of the Open-Label Extension Fixed Dose Phase
Description: Responders met the following criteria: >= 30%/50%/70% improvement in >= 3 of 6 JIA core criteria, and >= 30% worsening in not more than 1 JIA criterion, compared with OL baseline. JIA core criteria included: physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; # of active joints (joints with swelling or with LOM and with pain, tenderness or both); # of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein. Final Visit = last visit per subject (up to 224 weeks).
Time Frame: Final Visit (up to 224 weeks of OLE FD phase)
Population: The ITT population was used for analysis in the Open-Label Extension Fixed Dose phase.
Measure: Number; unit: Participants
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 55 | 46
Participants
  PedACR30 Final Visit | 48 | 44
  PedACR50 Final Visit | 45 | 43
  PedACR70 Final Visit | 43 | 40

19. Other Pre Specified Outcome: Baseline Measure: Gender, Female/Male - OLE BSA Phase
Description: Gender (female/male) recorded at Baseline of the Open-Label Extension BSA phase of the study. This measure was excluded from Baseline Characteristics due to difficulty maintaining correct subject numbers and Baseline value totals in that section while including this phase of the study.
Time Frame: Baseline OLE BSA Phase
Measure: Number; unit: Participants
Arm/Group | OLE BSA Adalimumab + MTX | OLE BSA Adalimumab
Number analyzed (Participants) | 71 | 57
Participants
  OLE BSA Phase - Female | 56 | 42
  OLE BSA Phase - Male | 15 | 15

20. Other Pre Specified Outcome: Baseline Measure: Age Continuous - OLE BSA Phase
Description: Age continuous (mean +/- SD) recorded at Baseline of the Open-Label Extension BSA phase of the study. This measure was excluded from Baseline Characteristics due to difficulty maintaining correct subject numbers and Baseline value totals in that section with this phase included.
Time Frame: Baseline OLE BSA Phase
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | OLE BSA Adalimumab + MTX | OLE BSA Adalimumab
Number analyzed (Participants) | 71 | 57
Years | 11.3 (3.32) | 11.2 (3.96)

21. Other Pre Specified Outcome: Baseline Measure: Gender, Female/Male - OLE FD Phase
Description: Gender (female/male) recorded at Baseline of the Open-Label Extension FD phase of the study. This measure was excluded from Baseline Characteristics due to difficulty maintaining correct subject numbers and Baseline value totals in that section while including this phase of the study.
Time Frame: Baseline OLE FD Phase
Measure: Number; unit: Participants
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 59 | 47
Participants
  OLE FD Phase - Female | 45 | 33
  OLE FD Phase - Male | 14 | 14

22. Other Pre Specified Outcome: Baseline Measure: Age Continuous - OLE FD Phase
Description: Age continuous (mean +/- SD) recorded at Baseline of the Open-Label Extension FD phase of the study. This measure was excluded from Baseline Characteristics due to difficulty maintaining correct subject numbers and Baseline value totals in that section with this phase included.
Time Frame: Baseline OLE FD Phase
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | OLE FD Adalimumab + MTX | OLE FD Adalimumab
Number analyzed (Participants) | 59 | 47
Years | 11.1 (3.36) | 11.0 (4.12)

ADVERSE EVENTS:
Time Frame: DB Phase - Week 16 to 48 (32 Weeks), Open-Label Extension BSA Phase - OLE BSA Baseline to Week 136 (136 weeks), Open-Label Extension FD Phase - OLE FD Baseline to Final Visit (up to 224 weeks)* *Last observation of each subject in FD population.
Groups:
- Open-Label Extension FD Adalimumab + MTX: Subjects in the methotrexate (MTX) stratum received adalimumab concomitantly with MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study, in which subjects were dosed based on body weight (not BSA). Subjects were separated into 2 body weight categories; subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
- Open-Label Extension FD Adalimumab: Subjects in the methotrexate (MTX) stratum received adalimumab without concomitant MTX treatment during the Open-Label Extension (OLE) Fixed Dose (FD) Phase of the study, in which subjects were dosed based on body weight (not BSA). Subjects were separated into 2 body weight categories; subjects weighing less than 30 kg were dosed with 20 mg of adalimumab SC eow, and subjects weighing 30 kg or more were dosed with 40 mg of adalimumab SC eow.
Arm/Group | Double-Blind Adalimumab + MTX | Double-Blind Placebo + MTX | Double-Blind Adalimumab | Double-Blind Placebo | Open-Label Extension BSA Adalimumab + MTX | Open-Label Extension BSA Adalimumab | Open-Label Extension FD Adalimumab + MTX | Open-Label Extension FD Adalimumab
Serious Adverse Events (participants affected / at risk) | 3/38 | 2/37 | 1/30 | 0/28 | 13/71 | 9/57 | 7/59 | 10/47
Other Adverse Events (participants affected / at risk) | 27/38 | 19/37 | 20/30 | 20/28 | 62/71 | 46/57 | 54/59 | 37/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Adalimumab + MTX (N=38) | Double-Blind Placebo + MTX (N=37) | Double-Blind Adalimumab (N=30) | Double-Blind Placebo (N=28) | Open-Label Extension BSA Adalimumab + MTX (N=71) | Open-Label Extension BSA Adalimumab (N=57) | Open-Label Extension FD Adalimumab + MTX (N=59) | Open-Label Extension FD Adalimumab (N=47)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 7
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Knee Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Adalimumab + MTX (N=38) | Double-Blind Placebo + MTX (N=37) | Double-Blind Adalimumab (N=30) | Double-Blind Placebo (N=28) | Open-Label Extension BSA Adalimumab + MTX (N=71) | Open-Label Extension BSA Adalimumab (N=57) | Open-Label Extension FD Adalimumab + MTX (N=59) | Open-Label Extension FD Adalimumab (N=47)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 2
Acute tonsillitis (Infections and infestations) | 1 | 2 | 0 | 0 | 4 | 0 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 5 | 6 | 4 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 4 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 5 | 2 | 2 | 4 | 3 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 6 | 5 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 1 | 7 | 4 | 2 | 4
Headache (Nervous system disorders) | 2 | 3 | 2 | 4 | 9 | 8 | 4 | 11
Herpes simplex (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 3
Impetigo (Infections and infestations) | 2 | 0 | 1 | 0 | 2 | 5 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 2 | 2 | 4 | 3 | 5
Influenza like illness (General disorders) | 0 | 4 | 0 | 0 | 4 | 1 | 0 | 0
Injection site burning (General disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 7 | 6 | 5 | 3 | 14 | 10 | 4 | 4
Injection site reaction (General disorders) | 7 | 1 | 3 | 1 | 8 | 9 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3 | 0 | 0 | 1 | 4
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 1 | 4 | 0 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 3 | 4 | 4
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 0 | 3 | 9 | 4 | 7 | 3
Pain (General disorders) | 1 | 1 | 3 | 3 | 0 | 3 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 1 | 9 | 4 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 1 | 4 | 6 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 5 | 4 | 2 | 6
Rhinitis (Infections and infestations) | 3 | 0 | 2 | 0 | 4 | 2 | 3 | 4
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 1 | 7 | 7 | 7 | 3
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 3
Thermal burn (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 6 | 5 | 21 | 19 | 15 | 13
Viral infection (Infections and infestations) | 6 | 2 | 6 | 3 | 13 | 9 | 15 | 8
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 5 | 3 | 2 | 3
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 9 | 3 | 2 | 6
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 6 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 4 | 5 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 7 | 7 | 7 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 4 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.